CLINICAL TRIAL: NCT03161041
Title: Perioperative Chemotherapy With Bevacizumab in Patients Undergoing Cytoreduction and Intraperitoneal Chemoperfusion for Colorectal Carcinomatosis - French Part of the Main Bev-IP Study
Brief Title: Perioperative Chemotherapy With Bevacizumab for Colorectal Carcinomatosis French Part of the Main Bev-IP Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: CHU Lyon will join as a participating center (and as national French coordinator) as a part of the BEV-IP study ongoing study EudraCT-number 2014-004257-14.
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL17_0239
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Colorectal Carcinomatosis
Keywords: Cytoreductive surgery, HIPEC, perioperative chemotherapy, peritoneal carcinomatosis, bevacizumab, colorectal surgery
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; Bevacizumab; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bevacizumab and CRS with oxaliplatin (Experimental): Perioperative chemotherapy plus bevacizumab and CRS with oxaliplatin
  Interventions: Procedure: Cytoreductive surgery combined with HIPEC; Drug: bevacizumab and HIPEC (Oxaliplatin 360 mg/m2).

INTERVENTIONS:
Procedure: Cytoreductive surgery combined with HIPEC — Procedure/Surgery: Cytoreductive surgery combined with HIPEC (Oxaliplatin 360 mg/m2).
Drug: bevacizumab and HIPEC (Oxaliplatin 360 mg/m2). — bevacizumab and HIPEC (Oxaliplatin 360 mg/m2).

SUMMARY:
Selected patients with peritoneal carcinomatosis (PC) from colorectal cancer (CRC) benefit from cytoreductive surgery (CRS) combined with intraperitoneal chemoperfusion (IPC). However, even after optimal cytoreduction, systemic and locoregional recurrence are common. Perioperative chemotherapy with bevacizumab (BEV) may improve the outcome of these patients. The BEV-IP study is a phase II, single-arm, open-label study aimed at patients with colorectal or appendiceal adenocarcinoma with synchronous or metachronous PC. This study evaluates whether perioperative chemotherapy including BEV in combination with CRS and oxaliplatin-based IPC results in acceptable morbidity and mortality (primary composite endpoint). Secondary endpoints are treatment completion rate, chemotherapy-related toxicity, pathological response, progression free survival, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* biopsy proven adenocarcinoma of the colon or rectum and synchronous or metachronous peritoneal carcinomatosis.
* absence of systemic disease, with the exception of small, superficial liver metastases, requiring only minor surgery.
* resectable disease at staging, during laparoscopic evaluation and during exploration for cytoreductive surgery and intraperitoneal chemotherapy.
* complete macroscopic cytoreduction at the time of surgery (CC-0/1)
* good general health status (Karnofsky index > 70%)
* expected life expectancy more than 6 months
* no other malignancy than disease under study
* serum creatinine < 1.5 mg/dl or a calculated GFR ≥ 60 mL/min/1.73 m2
* serum total bilirubin < 1.5 mg/dl
* platelet count > 100,000/ml
* hemoglobin > 9g/dl
* neutrophil granulocytes > 1,500/ml
* International Normalized Ration (INR) 2 or < 2
* Absence of alcohol and/or drug abuse
* No inclusion in other clinical trials interfering with the study protocol
* No concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy not indicated in the study protocol
* Absence of heart failure (NYHA 2 or > 2) or significant coronary artery disease
* No pregnancy or breast feeding
* Adequate contraception in fertile patients

Exclusion Criteria:

* No written informed consent
* Tumour in the presence of obstruction
* Evidence of extra-abdominal disease or extensive liver metastasis
* Peritoneal cancer index > 25
* Active bacterial, viral or fungal infection
* Active gastro-duodenal ulcer
* Parenchymal liver disease (any stage cirrhosis)
* Uncontrolled diabetes mellitus
* Severe obstructive or restrictive respiratory insufficiency
* Psychiatric pathology capable of affecting comprehension and judgment faculty
* Known allergy to oxaliplatin.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2018-11-13 (Estimated); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment related Adverse events grade IIIb or higher grade as assessed by Dindo-Clavien classification | Until 3 months after surgery and intraperitoneal chemotherapy
  Major morbidity (grade IIIb or higher grade complication according to Dindo-Clavien classification)

SECONDARY OUTCOMES:
Number of participants with treatement related Adverse events less than grade IIIb as assessed by Dindo-Clavien classification | Until 3 months after surgery and intraperitoneal chemotherapy
  Minor morbidity (less than grade IIIb complication according to Dindo-Clavien classification).
Potential chemotherapy related morbidity | During the first 60 postoperative days
  Adverse events will be described using MedDRA terms (version 18.0) and graded according to Common Terminology Criteria for Adverse Events (CTCAE version 5.0)
Overall survival | 24 months after finishing the adjuvant chemotherapy
  calculated from date of surgery until death
Progression free survival | 24 months after finishing the adjuvant chemotherapy
  Time interval between date of surgery and disease progression or death
Pathological gross response of peritoneal tumour deposits to neoadjuvant combination chemotherapy with bevacizumab | Day 1 after termination of the cytoreductive surgery
  Scored with a 3 level regression scale
Quality of life assessment | 24 months after finishing the adjuvant chemotherapy
  Using the EORTC QLQ-C30 questionnaires
Treatment completion rate | Day 1 after termination of adjuvant chemotherapy
  Percentage of patients receiving all planned courses
Quality of life assessment | 24 months after finishing the adjuvant chemotherapy
  Using SF 36 questionnaires

IPD SHARING:
Plan to Share IPD: No